CLINICAL TRIAL: NCT02837783
Title: A Phase 4, Single-centre, Randomised, Double-blind, Placebo-controlled, Parallel-group, Fixed-dose Study of the Effect of Linaclotide on Abdominal Girth in Participants With Irritable Bowel Syndrome With Constipation
Brief Title: A Study of the Effect of Linaclotide on Abdominal Girth in Participants With Irritable Bowel Syndrome With Constipation (IBS-C)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCP-103-403
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Irritable Bowel Syndrome Characterized by Constipation
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 290 μg linaclotide (Experimental): Linaclotide Oral, once daily
  Interventions: Drug: Linaclotide
- Matching Placebo (Placebo Comparator): Matching Placebo Oral, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linaclotide — Oral, once daily
  Arms: 290 μg linaclotide
Drug: Placebo — Oral, one daily
  Arms: Matching Placebo

SUMMARY:
The objective of this trial is to determine the effect of linaclotide on abdominal girth in IBS-C participants with the baseline symptoms of abdominal bloating and an increased abdominal girth.

ELIGIBILITY:
Inclusion Criteria:

• Patient meets protocol criteria for diagnosis of IBS-C, abdominal pain, abdominal bloating and abdominal girth

Exclusion Criteria:

* Patient has history of loose or watery stools
* Patient has both clinically significant findings and unexplained clinically significant alarm symptoms
* Patient has symptoms of or been diagnosed with a medical condition that may contribute to abdominal pain
* Patient has any protocol-excluded or clinically significant medical or surgical history that could confound the study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Whorwell, Principal Investigator — University Hospital of South Manchester
Locations (1):
- Peter Whorwell, Wythenshawe, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a 14-day screening period and a 7 day pretreatment period. The treatment period began with randomization and lasted for 4 weeks. Participants who met entry criteria were randomized (1:1) to once daily oral capsules containing 290 µg linaclotide or placebo.
Groups:
- Matching Placebo: Placebo once daily for 4 weeks
- 290 μg Linaclotide: 290 µg linaclotide once daily for 4 weeks
Period: Overall Study
Arm/Group | Matching Placebo | 290 μg Linaclotide
Started | 9 | 11
Received >= 1 Dose of Study Drug | 9 | 10
Completed | 7 | 9
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Other, Not Specified | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- 290 μg Linaclotide: 290 μg linaclotide once daily for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Matching Placebo | 290 μg Linaclotide | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (10.38) | 35.2 (12.82) | 35.5 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 9 | 11 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Abdominal Girth at Week 4
Description: Mean change in abdominal girth (physical measure of bloating/distension) as measured by area under the curve (AUC), determined by 24-hour abdominal inductance plesthymography (AIP; with hourly averages). The AUC was calculated using the Trapezoidal method from the first reliable hour of measurement to last measurement (bedtime). The AUC for each participant was then individually standardized by dividing the total AUC over the period by that patient's number of hours of measurement included in the AUC. (Therefore, the time element was removed from the standardized AUC, and the unit of measure for this outcome is centimeters [cm]).
Time Frame: Baseline, Week 4
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Matching Placebo | 290 μg Linaclotide
Number analyzed (Participants) | 9 | 11
cm
  Baseline | 82.6 (11.8) | 83.7 (9.02)
  Change From Baseline: number analyzed (Participants) | 7 | 10
  Change From Baseline | -3.36 (4.04) | -0.632 (11.6)
Statistical Analysis 1: Comparison: Matching Placebo vs 290 μg Linaclotide; Test type: Superiority; p = 0.283, Wilcoxon rank sum test

2. Secondary Outcome: Change From Baseline in Abdominal Girth at Week 2
Description: Mean change in abdominal girth (physical measure of bloating/distention) as measured by AUC, determined by 24-hour AIP (with hourly averages). The AUC was calculated using the Trapezoidal method from the first reliable hour of measurement to last measurement (bedtime). The AUC for each participant was then individually standardized by dividing the total AUC over the period by that patient's number of hours of measurement included in the AUC. (Therefore, the time element was removed from the standardized AUC, and the unit of measure for this outcome is centimeters [cm]).
Time Frame: Baseline, Week 2
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Matching Placebo | 290 μg Linaclotide
Number analyzed (Participants) | 8 | 10
cm | 0.535 (9.15) | -2.3 (13.7)

3. Secondary Outcome: Percent Change From Baseline in Maximal Abdominal Girth at Week 4
Description: The maximum change in girth from the first hour, over the period from the 2nd hour to bedtime. The percentage change in maximum distension from baseline to 4 weeks will also be calculated.
Time Frame: Baseline, Week 4
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Matching Placebo | 290 μg Linaclotide
Number analyzed (Participants) | 7 | 9
percent change | -7.13 (33.4) | 15.4 (80.3)

4. Secondary Outcome: Change From Baseline of Symptom Severity (Abdominal Pain, Discomfort, Bloating, and Distension) at Week 1
Description: Symptom severity was assessed daily on an 11-point numerical rating scale (NRS) from 0 to 10, where 0 represents no symptoms and 10 represents very severe symptoms. Participants rated their abdominal pain, discomfort, bloating, and distension at its worst over the last 24 hours. Weekly average scores were calculated individually for abdominal pain, discomfort, bloating, distension. The abdominal score was calculated as the weekly average from the daily scores of the individual items of pain, discomfort, bloating combined. The abdominal score plus distension was calculated as the weekly average from the daily scores of the individual items of pain, discomfort, bloating and distension combined.
Time Frame: Baseline, Week 1
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Matching Placebo | 290 μg Linaclotide
Number analyzed (Participants) | 8 | 11
units on a scale
  Pain | -1.25 (1.76) | -0.75 (1.88)
  Discomfort | -1.93 (1.54) | -0.97 (2.05)
  Bloating | -2.00 (1.48) | -0.40 (1.23)
  Distension | -1.91 (1.41) | -0.15 (1.02)
  Abdominal Score | -1.73 (1.50) | -0.71 (1.58)
  Abdominal Score + Distension | -1.77 (1.43) | -0.57 (1.36)

5. Secondary Outcome: Change From Baseline of Symptom Severity (Abdominal Pain, Discomfort, Bloating, and Distension) at Week 2
Description: Symptom severity was assessed daily on an 11-point NRS from 0 to 10, where 0 represents no symptoms and 10 represents very severe symptoms. Participants rated their abdominal pain, discomfort, bloating, and distension at its worst over the last 24 hours. Weekly average scores were calculated individually for abdominal pain, discomfort, bloating, distension. The abdominal score was calculated as the weekly average from the daily scores of the individual items of pain, discomfort, bloating combined. The abdominal score plus distension was calculated as the weekly average from the daily scores of the individual items of pain, discomfort, bloating and distension combined.
Time Frame: Baseline, Week 2
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Matching Placebo | 290 μg Linaclotide
Number analyzed (Participants) | 8 | 10
units on a scale
  Pain | -1.97 (1.60) | -1.42 (1.88)
  Discomfort | -2.51 (1.15) | -1.73 (2.27)
  Bloating | -2.65 (1.30) | -1.04 (1.54)
  Distension | -2.51 (1.37) | -0.78 (1.33)
  Abdominal Score | -2.38 (1.19) | -1.40 (1.69)
  Abdominal Score + Distension | -2.41 (1.18) | -1.25 (1.52)

6. Secondary Outcome: Change From Baseline of Symptom Severity (Abdominal Pain, Discomfort, Bloating, and Distension) at Week 3
Description: as for outcome 5
Time Frame: Baseline, Week 3
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Matching Placebo | 290 μg Linaclotide
Number analyzed (Participants) | 8 | 10
units on a scale
  Pain | -1.60 (2.66) | -2.07 (1.88)
  Discomfort | -2.01 (1.86) | -2.25 (2.26)
  Bloating | -2.02 (1.67) | -1.16 (1.51)
  Distension | -1.79 (1.80) | -1.05 (1.37)
  Abdominal Score | -1.88 (1.95) | -1.82 (1.64)
  Abdominal Score + Distension | -1.86 (1.87) | -1.64 (1.46)

7. Secondary Outcome: Change From Baseline of Symptom Severity (Abdominal Pain, Discomfort, Bloating, and Distension) at Week 4
Description: as for outcome 5
Time Frame: Baseline, Week 4
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Matching Placebo | 290 μg Linaclotide
Number analyzed (Participants) | 8 | 10
units on a scale
  Pain | -1.71 (2.44) | -1.90 (1.50)
  Discomfort | -1.94 (1.63) | -2.24 (1.92)
  Bloating | -1.84 (1.64) | -1.64 (1.74)
  Distension | -1.70 (1.60) | -1.22 (1.69)
  Abdominal Score | -1.83 (1.84) | -1.91 (1.39)
  Abdominal Score + Distension | -1.80 (1.75) | -1.74 (1.37)

8. Secondary Outcome: Change From Baseline in Digestive Sensations (Subjective Bloating, Abdominal Discomfort, Abdominal Distension and Abdominal Pain) at Week 2
Description: A digestive sensations questionnaire was used to record abdominal pain, discomfort, bloating, and distension symptoms on an hourly basis (waking hours only) during the 24 hours the participants are fitted with the AIP belt, using an 11-point NRS, with 0=no symptomatic sensations and 10=most severe symptomatic sensations. Daily diary scores for each of the digestive symptoms was averaged to obtain 'weekly' scores.
Time Frame: Baseline, Week 2
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Matching Placebo | 290 μg Linaclotide
Number analyzed (Participants) | 8 | 10
units on a scale
  Pain | -1.13 (1.38) | -0.61 (1.10)
  Discomfort | -1.01 (1.53) | -1.00 (1.34)
  Bloating | -1.03 (1.54) | -0.58 (1.33)
  Distension | -0.97 (1.50) | -0.36 (1.14)

9. Secondary Outcome: Change From Baseline in Digestive Sensations (Subjective Bloating, Abdominal Discomfort, Abdominal Distension and Abdominal Pain) at Week 4
Description: A digestive sensations questionnaire was used to record abdominal pain, discomfort, bloating, and distension on an hourly basis (waking hours only) during the 24 hours the participants are fitted with the AIP belt, using an 11-point NRS, with 0=no symptomatic sensations and 10=most severe symptomatic sensations. Daily diary scores for each of the digestive symptoms was averaged to obtain 'weekly' scores.
Time Frame: Baseline, Week 4
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Matching Placebo | 290 μg Linaclotide
Number analyzed (Participants) | 7 | 9
units on a scale
  Pain | -0.97 (1.55) | -0.87 (1.33)
  Discomfort | -0.89 (1.51) | -1.81 (1.11)
  Bloating | -1.01 (1.57) | -1.66 (1.03)
  Distension | -1.03 (1.49) | -1.42 (0.64)

10. Secondary Outcome: Change From Baseline in Bristol Stool Form Scale (BSFS) Over Time
Description: Daily stool consistency analyses were performed using the 7-point Bristol Stool Form Scale (BSFS), whereby a score of 1 = separate hard lumps like nuts (difficult to pass); 2 = sausage shaped but lumpy; 3 = like a sausage but with cracks on surface; 4 = like a sausage or snake, smooth and soft; 5 = soft blobs with clear-cut edges (passed easily); 6 = fluffy pieces with ragged edges, a mushy stool; and 7 = watery, no solid pieces (entirely liquid). Daily average recorded BSFS scores for each participant were computed for each week.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4
Population: Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Matching Placebo | 290 μg Linaclotide
Number analyzed (Participants) | 8 | 11
score on a scale
  Week 1 | 0.33 (0.88) | 1.53 (1.57)
  Week 2: number analyzed (Participants) | 8 | 10
  Week 2 | 0.57 (0.86) | 1.51 (1.27)
  Week 3: number analyzed (Participants) | 8 | 10
  Week 3 | 0.39 (1.15) | 2.11 (1.43)
  Week 4: number analyzed (Participants) | 8 | 10
  Week 4 | 0.35 (1.11) | 1.56 (1.13)

ADVERSE EVENTS:
Time Frame: From first dose of study drug through Day 36 (± 2 days).
Arm/Group | Matching Placebo | 290 μg Linaclotide
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/10
Other Adverse Events (participants affected / at risk) | 1/9 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Matching Placebo (N=9) | 290 μg Linaclotide (N=10)
Loss of consciousness (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Matching Placebo (N=9) | 290 μg Linaclotide (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 5
Nausea (Gastrointestinal disorders) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to an insufficient sample size, no conclusions could be drawn regarding efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (2):
  • Study Protocol (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT02837783/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT02837783/SAP_001.pdf